CLINICAL TRIAL: NCT06288464
Title: Does Distal Enteral Feeding of Fibre Positively Affect the Microflora in the Distal Limb of Loop Ileostomy Patients?
Brief Title: Enteral Feeding of Fibre to Improve Microbiota
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lancashire Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Lancaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 315656; 22/WM/0222 (Other: Health Research Authority)
Record Dates: First submitted 2024-02-09; First posted 2024-03-01 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Bowel Dysfunction; Colon Disease; Ileum--Diseases
MeSH Terms: conditions — Intestinal Diseases; Colonic Diseases

STUDY DESIGN:
Intervention Model Description: Cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Stoma feeding
  Interventions: Dietary Supplement: Soluble Fibre

INTERVENTIONS:
Dietary Supplement: Soluble Fibre — Patients will be assigned to stoma feeding by the Colorectal Surgeon, which will be managed by the stoma nurses for the duration, approximately 4 weeks, of feeding. For the final 7-14 days (minimum 7 days) of feeding, 10g of soluble fibre will be added to 100ml of Ensure™ (or equivalent liquid nutrient feed) before instillation into the stoma on a daily basis. The soluble fibre will be provided in 10g portions and should be added to the newly-opened bottle of ensure and shaken to mix well.

SUMMARY:
Following surgical removal of diseased bowel, patients often require a temporary redirection of bowel contents to a stoma, to allow healing prior to re-joining of the remaining bowel at a later date. Some patients may experience complications, either during or after reversal surgery, and this may be due to changes in the 'friendly' bacteria that live in our bowels. Previous research shows that the distal section of bowel that is non-functioning undergoes tissue-wasting and the 'friendly' bacteria that help our digestion die. Data shows that patients that have a reduction in their microflora are more likely to experience side effects. This study investigates a method of replenishing the microflora prior to surgery.

DETAILED DESCRIPTION:
Surgical formation of a loop ileostomy to divert the faecal stream and allow tissue healing, with the aim of re-joining the bowel around 1 year later, is carried out in around 9000 patient per year in the United Kingdom (UK). One in 4 patients experience severe side effects, such as inflammation or lack of function following reversal, and 5% of patients cannot undergo reversal, leaving them with a permanent stoma. Previous data shows that patients with less bacteria in the distal bowel may be more likely to develop post-operative complications. This study investigates a method of replenishing the microflora prior to surgery. The data also shows that patients with less bacteria in the distal bowel may be more likely to develop post-operative complications.

This study will pilot a clinical trial to assess whether enteral feeding in these 'high risk' patients alters the microflora, prior to applying to complete a randomised, controlled trial to assess the effectiveness of enteral feeding in standard-care patients. The enteral feeding is carried out through a feeding tube into the defunctioned part of the stoma. Initially patients receive saline and build up to approximately 100ml of 'Ensure™', a nutrition shake containing 9 amino acids and various vitamins and minerals, over a period of approximately 4 weeks. A source of fibre will be added to the shake, a Chicory root extract made by BENEO™, for the final week to 10 days of stoma feeding. There is evidence to support that oral consumption, in both adult and paediatric patients, of the chicory root extract supports positive microflora growth. We propose to supplement Ensure™ with up to 10g of chicory root extract for the final 7-10 days of stoma feeding and assess the changes on both the microbiota and on the histological and biomolecular properties of the intestinal tissues.

This research aims to investigate ways to increase the numbers of friendly bacteria to improve the health of the distal, non-functioning, bowel by adding fibre to the nutritional supplement fed to the distal bowel for around two weeks prior to surgery. The aim is that this will reduce the risk of complications and possibly reduce the recovery time from bowel surgery.

ELIGIBILITY:
Inclusion Criteria:

* Any individual that has been identified for distal (stoma) feeding that is able to understand verbal and written English to provide informed consent.
* Participants must be undergoing ileostomy or colostomy reversal surgery.

Exclusion Criteria:

* Not undergoing ileostomy or colostomy reversal.
* Persons who might not adequately understand verbal explanations or written information given in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of Microbiota | 1 month
  16S rRNA sequencing and qPCR, comparing de-functioned and functional limbs of the ileostomy.
  Biomolecular analysis of the tissues, to assess growth and inflammation, using histological techniques to quantify and identify the microbiota.
Concentration of Immune Cell Populations | 1 month
  Immune cell populations will be identified and profiled using flow cytometric analysis and/or immunohistochemistry.

SECONDARY OUTCOMES:
Length of Stay | 1 month
  Length of stay in hospital
Rate of clinical complications | 1 month
  Clinical observations or complications (e.g. anastomotic leak, ileus, excessive distention/bloating or wound infection) will be recorded.
  Along with information regarding Patient BMI, sex, date of stoma creation, and history of antibiotic usage (name/duration) during the time stoma was in place should also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Kina Bennett, Study Chair — Lancashire Teaching Hospitals NHS Foundation Trust
Locations (1):
- Lancashire Teaching Hospitals NHS, Preston, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT06288464/Prot_000.pdf